CLINICAL TRIAL: NCT00854464
Title: Arsenic Methylation, Cigarette Smoking Exposure, Individual DNA Susceptibility Factors and Urothelial Carcinoma
Brief Title: Arsenic Methylation Enzymes, Cigarette Metabolites, DNA Repair Enzymes, Inflammatory Factors and Urothelial Carcinoma
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Yeong-Shiau Pu, Department of Urology / National Taiwan University Hospital
Other Study IDs: 200809019R
Record Dates: First submitted 2009-03-01; First posted 2009-03-03 (Estimated); Last update posted 2009-03-03 (Estimated); Status verified 2009-03

CONDITIONS: Urothelial Carcinoma
Keywords: Arsenic Methylation Capability; Arsenic Methylation Enzymes; Cigarette Metabolites; Cigarette Metabolic Enzymes; DNA Repair Enzymes; Inflammatory Factors; Urothelial Carcinoma
MeSH Terms: conditions — Carcinoma, Transitional Cell

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

SUMMARY:
1. To investigate the relationship between arsenic methylation enzymes (AS3MT, PNP,GSTO1, and GSTO2) genetic polymorphism and UC risk.
2. To explore the relationship between cigarettes metabolites (NNK, NNAL, HBA, NNAL-Gluc, O6-Methylguanine, and N7-Methylguanine) and UC risk.
3. To examine the relationship between cigarette metabolic enzymes (CYP2A6, CYP2A13, and UGT2B7) genetic polymorphism and UC risk.
4. To elucidate the relationship between DNA repair enzymes (MGMT, XPD, XRCC1, and XRCC3) gene polymorphism and 8-OHdG or between DNA repair enzymes and UC risk.
5. To examine relationship between COX-2 (-1195G/A、-765G/C 和8473C/T), IL-6, IL-8, and TNF-α gene polymorphism and 8-OHdG or between COX-2, IL-6, IL-8, and TNF-α gene polymorphism and UC risk.
6. To examine the risk factors of the environment-environment, gene-environment, and gene-gene interaction on the risk of UC.

DETAILED DESCRIPTION:
Urothelial carcinoma (UC) arises exclusively from the urothelium including the renal pelvis,ureter, bladder and urethra, with bladder transitional cell carcinoma (TCC) being the most common form. Arsenic is a well-established human carcinogen of the skin and lung. Recent studies have well documented that the long-term exposure to inorganic arsenic through ingestion and inhalation is associated with an increased risk of bladder cancer, especially TCC.

However, the carcinogenic mechanism of arsenic-induced UC is still unclear. Recently our study found that cigarette smoking interacts with the urinary arsenic profile in modifying the UC risk. In addition, we also found that DNA damage marker 8-hydroxydeoxyguanine (8-OHdG) levels significantly higher in UC patients compared to healthy controls. The mechanism of the interaction between arsenic methylation and cigarette on UC risk is unknown. In addition, whether 8-OHdG is related to DNA repair enzymes or to inflammatory factors or not does need to explore, therefore the specific aims of this project are:

1. To investigate the relationship between arsenic methylation enzymes (AS3MT, PNP, GSTO1, and GSTO2) genetic polymorphism and UC risk.
2. To explore the relationship between cigarettes metabolites (NNK, NNAL, HBA, NNAL-Gluc, O6-Methylguanine, and N7-Methylguanine) and UC risk.
3. To examine the relationship between cigarette metabolic enzymes (CYP2A6, CYP2A13, and UGT2B7) genetic polymorphism and UC risk.
4. To elucidate the relationship between DNA repair enzymes (MGMT, XPD, XRCC1, and XRCC3) gene polymorphism and 8-OHdG or between DNA repair enzymes and UC risk.
5. To examine relationship between COX-2 (-1195G/A、-765G/C 和8473C/T), IL-6, IL-8, and TNF-α gene polymorphism and 8-OHdG or between COX-2, IL-6, IL-8, and TNF-α gene polymorphism and UC risk.
6. To examine the risk factors of the environment-environment, gene-environment, and gene-gene interaction on the risk of UC.

ELIGIBILITY:
Inclusion Criteria:

* project recruited 420 UC patients in Taiwan University Hospital

Exclusion Criteria:

-

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: project recruited 420 UC patients in Taiwan University Hospital
Sampling Method: Non-Probability Sample
Enrollment: 420 (Estimated)
Dates: Start 2008-08; Primary Completion 2011-07 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Yeong-Shiau Pu, M.D.PhD., Principal Investigator — National Taiwan University Hospital
Locations (1):
- Department of Urology/National Taiwan University Hospital, Taipei, Taiwan